CLINICAL TRIAL: NCT05128929
Title: Investigation of H01 in Adults With Pulmonary Hypertension Including Interstitial Lung Disease (The SATURN Study).
Acronym: SATURN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Roham T. Zamanian, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H01
Record Dates: First submitted 2021-11-11; First posted 2021-11-22 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Hypertension
Keywords: Six Minute Walk Distance Test (6 MWDT); Right Heart Catheterization (RHC); Pulmonary Vascular Resistance (PVR); Pulmonary Function Test (PFT); Mean Pulmonary Arterial Pressure (mPAP); Pharmacokinetics; Pharmacodynamics; Hyaluronan; Hymecromone
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Hymecromone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment Oral Hymecromone (H01) (Experimental): Treatment will be initiated. Participants will be administered 800 mg of oral H01 two times a day (total dose: 1600 mg/day). Participants will continue to be on treatment for 24 weeks and will be monitored with assessments.
  Interventions: Drug: Hymecromone (H01)
- Placebo (Placebo Comparator): Participants randomized to placebo will receive oral tablet placebo (inactive ingredients) two times a day. Participants will continue to be on placebo for 24 weeks and will be monitored with assessments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hymecromone (H01) — 800 mg oral H01 two times a day (total dose: 1600 mg/day).
  Other Names: Cantabiline; Isochol
  Arms: Experimental Treatment Oral Hymecromone (H01)
Drug: Placebo — Oral tablet placebo (inactive ingredients) two times a day.
  Arms: Placebo

SUMMARY:
This study is a prospective, randomized, double-blind, study of H01 (Hymecromone) in adults with pulmonary hypertension (PH). The primary objective of this study is to evaluate the safety and tolerability of oral H01 and the potential benefit of oral H01 on clinical measures of PH disease severity over 24 weeks.

Study Hypothesis:

Oral H01, at doses of 1600 mg per day, will be a safe and well-tolerated agent in adults with pulmonary hypertension over 24 weeks

DETAILED DESCRIPTION:
The study's objectives are to evaluate:

* The changes in clinical and functional measures (pulmonary function test, pulmonary vascular resistance, mean pulmonary arterial pressure, and 6 Minute Walk Distance Test) in adults with PH treated with oral H01
* The safety and tolerability of the use of oral H01 for PH over 24 weeks using health criteria/evaluations (Common Terminology Criteria for Adverse Events (CTCAE), quality of life (QOL) score, EMPHASIS-10 score and St George Respiratory Questionnaire (SGRQ) score)
* To investigate the clinical efficacy, pharmacokinetic (PK) and pharmacodynamic (PD) markers (serum HA concentration, inflammatory markers and cytokines, NT-proBNP, and H01 and metabolite serum concentrations) in this population following oral H01 use

ELIGIBILITY:
Inclusion Criteria:

1. Classified as WHO functional class II/III/IV despite treatment with maximally tolerated doses of 2 or more treatment modalities (exp. PDE5 inhibitors, guanylate cyclase stimulators, endothelin receptor antagonists, and prostanoids)
2. Baseline 6MWT: greater than 100 meters and less than 550 meters
3. Established diagnosis of Group 3 pulmonary hypertension as a result of interstitial lung disease OR established diagnosis of Group 1 pulmonary hypertension as a result of connective tissue disease, idiopathic, hereditary, drugs, or toxins.
4. Right heart catheterization at randomization showing pre-capillary pulmonary hypertension (mPAP ≥ 25 mmHg and PVR > 400 dynes * sec * cm^ -5) and:

   * PCWP ≤20 mmHg for Group 3 PH patients and Group 1 PAH patients
5. Participants on chronic medication for PAH, PH, or underlying lung disease must be on a stable and optimized dose for at least 90 days prior to the first dose of the study drug.
6. Female participants who are heterosexually active must use an acceptable method of contraception: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, IUD, or Hormone-based contraceptive
7. Be able to provide written informed consent and comply with study requirements
8. Be able to read, speak and understand English

Exclusion Criteria:

1. Participants with a diagnosis of PAH or PH for reasons due to any of the following:

   * Group 2, 4, or 5
   * Group 1 due to HIV, veno-occlusive disease, porto-pulmonary hypertension, congenital heart disease
   * Group 3 due to severe chronic obstructive pulmonary disease (COPD) or obstructive sleep apnea (OSA)

     * Note: participants with overlapping syndromes will be evaluated on a case-by-case basis by the recruiting physician*
2. Total Lung Capacity (TLC) less than 60% predicted
3. FEV1/FVC less than 50% predicted or FEV1 less than 55% predicted
4. Inability to safely attempt completion of the 6MWD test
5. Use of experimental PAH treatments within the past 3 months
6. Current systemic treatment with hymecromone
7. Left sided heart disease as defined by either a PCWP greater than 20 mmHg and/or left ventricular ejection fraction less than 40%

   * Note: participants with abnormal left ventricular function attributable entirely to impaired left ventricular filling due to the effects of right ventricular overload (ie right ventricular hypertrophy and/or dilatation) are not excluded
8. Participants must not have 3 or more of the following left ventricular disease / dysfunction risk factors:

   * Body mass index (BMI) greater than 30kg/m2
   * History of essential hypertension requiring medication
   * Diabetes mellitus
9. Historical evidence of significant coronary disease established by any of the following:

   * History of myocardial infarction
   * History of percutaneous coronary intervention or coronary artery bypass graft
   * Angiographic evidence of greater than 50% stenosis in at least one coronary artery
   * Positive stress test with imaging
   * Stable angina
10. Significant valvular heart disease as determined by more than moderate findings on echocardiogram or history of valve replacement
11. Pregnant or actively breastfeeding
12. Female participants with childbearing potential not willing to use a form of birth control (including abstinence) during the study
13. Inability to undergo right heart catheterization
14. Acute pulmonary embolism within 90 days of randomization
15. Exacerbation of underlying lung disease or active pulmonary or upper respiratory infection within 30 days of randomizations
16. Use of any inhaled tobacco products or significant history of drug abuse within 3 months prior to randomization
17. Subject is receiving greater than 10L/min of oxygen supplementation by any mode of delivery at rest at baseline
18. Body mass index greater than 40kg/m2
19. Participants with history of dysphagia, achalasia, or difficulty swallowing capsules, tablets or pills
20. Participants with liver failure or AST or ALT greater than 2 times the upper limit of normal
21. Participants with total bilirubin levels greater than 2 times the upper limit of normal
22. Participants with CrCl less than 45
23. Use of any investigational drug/device, or participation in any investigational study with therapeutic intent within 30 days prior to randomization
24. Known allergy to hymecromone or any component thereof
25. Known allergy to any component of placebo (including wheat allergy, celiac disease, rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption)
26. Physician concern that participant may not adhere to the study protocol
27. Significant psychiatric, addictive, or other disorder that compromises the subject's ability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Czepiel K, Nagy N, Panjalingam T, Kalinowski A, Frymoyer AR, Karmouty-Quintana H, Gu B, Hedlin H, Kaber G, Dobrota Lai S, Rosser JI, Bollyky PL, de Jesus Perez V, Zamanian RT. Randomised, placebo-controlled trial of oral hymecromone in adults with pulmonary hypertension. Thorax. 2025 Aug 15;80(9):632-640. doi: 10.1136/thorax-2024-222725. PMID 40451287
- [Derived] Salman L, Martinez L, Faddoul G, Manning C, Ali K, Salman M, Vazquez-Padron R. Hyaluronan Inhibition as a Therapeutic Target for Diabetic Kidney Disease: What Is Next? Kidney360. 2023 Jun 1;4(6):e851-e860. doi: 10.34067/KID.0000000000000126. Epub 2023 Apr 14. PMID 37055910

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants signed the informed consent. Out of these 17 participants,16 were randomized and started the study. The planned open-label extension study did not occur.
Groups:
- Experimental Treatment Oral Hymecromone (H01): Participants receive H01 800 mg oral H01 two times a day (total dose: 1600 mg/day).
- Placebo: Participants receive oral tablet placebo (inactive ingredients) two times a day.
Period: Overall Study
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Started | 10 | 6
Primary Analysis (Week 24) | 10 | 6
Completed | 10 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (12.4) | 66.5 (3.73) | 58.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Calculated Pulmonary Vascular Resistance (PVR)
Description: Calculated pulmonary vascular resistance (PVR) measured by right heart catheterization (RHC).
  A normal PVR ranges between 0.25 and 1.6 wood units (WU). Pre-capillary pulmonary hypertension is characterized by a PVR greater than 3 WU. Greater PVR is indicative of increased disease severity.
  Either Fick or Thermodilution method can be utilized to measure cardiac output (CO) and calculate PVR. Fick method utilizes estimated oxygen consumption to measure CO and calculate PVR, while the thermodilution method utilizes temperature change to measure CO and calculate PVR.
  All measurements to calculate PVR were obtained at end-expiration (measuring the pressures at functional residual capacity of the lungs).
Time Frame: Baseline to end of treatment (Week 24; +/- 7 days)
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: Wood units (WU)
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
Wood units (WU)
  Baseline - TD method | 7.97 (2.65) | 8.23 (4.16)
  Week 24 - TD method: number analyzed (Participants) | 10 | 5
  Week 24 - TD method | 7.27 (2.83) | 7.11 (2.69)
  Baseline - Fick method | 9.04 (3.52) | 9.97 (5.84)
  Week 24 - Fick method: number analyzed (Participants) | 10 | 5
  Week 24 - Fick method | 9.14 (3.39) | 8.03 (1.10)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; Null: There is no significant difference in the mean primary endpoint (PVR) at 24 weeks between the treatment (H01) and placebo group. The following analysis utilizes PVR determined by TD; Test type: Superiority; p = 0.541, Mixed Models Analysis; Analysis was adjusted for the randomization stratum of PAH Group; Mean Difference (Final Values) = 0.614, 95% CI 2-sided [-1.47 to 2.79]

2. Secondary Outcome: Number of Participants With Adverse Events by Severity Using the NIH Common Terminology Criteria for Adverse Events (CTCAE) as a Measure of Safety and Tolerability of H01 in Adults With Pulmonary Hypertension
Description: * Grade 1: Mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2: Moderate minimal, local or noninvasive intervention indicated; limiting age- appropriate instrumental activities of daily living (ADL).
  * Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
  * Grade 4: Life-threatening consequences; urgent intervention indicated.
  * Grade 5: Death related to AE.
Time Frame: Baseline to end of treatment (Week 24; +/- 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
Participants
  Grade 1 (mild) | 3 | 1
  Grade 2 (moderate) | 1 | 3
  Grade 3 (severe) | 0 | 2
  Grade 4 (life-threatening) | 0 | 0
  Grade 5 (death) | 0 | 0

3. Secondary Outcome: Mean Pulmonary Arterial Pressure (mPAP)
Description: Mean pulmonary arterial pressure (mPAP) measured by RHC.
  A normal mPAP ranges between 9 and 19 mmHg at rest. Pre-capillary pulmonary hypertension is characterized by a mPAP greater than 20 mmHg at rest. Greater mPAP is indicative of increased disease severity.
  All measurements were obtained at end-expiration.
Time Frame: Baseline and end of treatment (Week 24; +/- 7 days)
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
mmHg
  Baseline | 43.6 (10.0) | 47.5 (9.40)
  Week 24: number analyzed (Participants) | 10 | 5
  Week 24 | 40.2 (10.9) | 42.4 (9.34)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; Null: There is no significant difference in the mean secondary endpoint (mPAP) at 24 weeks between the treatment (H01) and placebo group; Test type: Superiority; p = 0.599, Mixed Models Analysis; Analysis was adjusted for the randomization stratum of PAH Group; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [-4.34 to 7.27]

4. Secondary Outcome: 6 Minute Walk Distance Test (6 MWDT)
Description: The 6MWDT (distance walked in 6 minutes) is used to determine functional exercise capacity, assess treatment efficacy, predict prognosis, and establish rehabilitation programs in PAH/PH patients.
Time Frame: Screening (up to 30 days prior to baseline) and weeks 4 (+/- 3 days), 12 (+/- 3 days), and 24 (+/- 7 days).
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
meters
  Screening | 409.0 (110.0) | 355.0 (73.5)
  Week 4 | 383.0 (104.0) | 347.0 (92.1)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | 441.0 (91.1) | 361.0 (127.0)
  Week 24 | 429.0 (101.0) | 340.0 (112.0)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; Null: There is no significant difference in the mean secondary endpoint (6MWT distance) at 24 weeks between the treatment (H01) and placebo group; Test type: Superiority; p = 0.166, Mixed Models Analysis; Analysis was adjusted for the randomization stratum of PAH Group; Mean Difference (Final Values) = 47.26, 95% CI 2-sided [-21.43 to 115.95]

5. Secondary Outcome: EMPHASIS-10 Scale Score
Description: Quality of life (QOL) assessed using the EMPHASIS-10 questionnaire.
  The minimum score for this questionnaire is 0. The maximum score for this questionnaire is 50. Higher scores are indicative of poorer health-related quality of life (HRQoL) due to pulmonary hypertension.
Time Frame: Baseline and weeks 4 (+/- 3 days), 12 (+/- 3 days), and 24 (+/- 7 days)
Population: Participants with data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
score on a scale
  Baseline | 20.6 (9.9) | 19.3 (12.0)
  Week 4 | 22.1 (9.6) | 19.8 (12.2)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | 19.0 (7.8) | 15.0 (12.3)
  Week 24 | 15.0 (7.6) | 14.3 (10.5)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; Null: There is no significant difference in the mean secondary endpoint (emPHasis-10 score) at 24 weeks between the treatment (H01) and placebo group; Test type: Superiority; p = 0.975, Mixed Models Analysis; Analysis was adjusted for the randomization stratum of PAH Group; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-8.22 to 7.98]

6. Secondary Outcome: St George Respiratory Questionnaire (SGRQ) Scale Score
Description: Quality of life (QOL) assessed using the St George Respiratory Questionnaire (SGRQ).
  There are a total of 3 components in the questionnaire, including symptoms, activity, and impacts. Each component has a minimum weight of 0, and a maximum weight of 662.5, 1209.1, and 2117.8, respectively. The minimum weight of the total score (combining all 3 components) is 0, and the maximum weight of total score is 3989.4.
  The total score is calculated by dividing the summed weights from positive items in the questionnaire by the sum of weights for all items in the questionnaire and multiplying this by 100. The minimum total score is 0, the maximum is 100.
  Lower scores indicate better health status.
Time Frame: Baseline and weeks 4 (+/- 3 days), 12 (+/- 3 days), and 24 (+/- 7 days)
Population: Participants with data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
score on a scale
  Baseline | 32.9 (13.3) | 36.0 (17.4)
  Week 4 | 38.1 (15.4) | 35.2 (19.2)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | 31.0 (9.42) | 36.5 (23.9)
  Week 24 | 27.8 (9.88) | 39.1 (27.1)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; Null: There is no significant difference in the mean secondary endpoint (SGRQ Score) at 24 weeks between the treatment (H01) and placebo group; Test type: Superiority; p = 0.086, Mixed Models Analysis; Analysis was adjusted for the randomization stratum of PAH Group; Mean Difference (Final Values) = -9.00, 95% CI 2-sided [-19.40 to 1.4]

7. Secondary Outcome: Serum Hyaluronan (HA) Concentration
Description: Two samples were collected at each time point and mean values were calculated. The average of the two mean values is reported.
  The normal adult circulating level of hyaluronan ranges between 10 and 100 ng/mL.
Time Frame: Baseline and end of treatment (Week 24; +/- 7 days)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
ng/mL
  Baseline | 181 (70) | 186 (32.8)
  Week 24 | 222 (193) | 149 (39.6)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; Null: There is no significant difference in the mean secondary endpoint (serum HA) at 24 weeks between the treatment (H01) and placebo group; Test type: Superiority; p = 0.215, Mixed Models Analysis; Analysis was adjusted for the randomization stratum of PAH Group; Mean Difference (Final Values) = 73.92, 95% CI 2-sided [-45.61 to 193.46]

8. Secondary Outcome: N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: N-terminal pro-brain-type natriuretic peptide (NT-proBNP) is laboratory test used for assessing disease severity in pulmonary hypertension.
  The normal ranges for NT-proBNP are as follows:
  Male (Reflects 95th percentile w/o CHF ):
  18-<44 yr: 36-93 pg/mL 44-<54 yr: 36-138 pg/mL 54-<64 yr: 36-177 pg/mL 64-<74 yr: 36-229 pg/mL 74 yr: 36-852 pg/mL
  Females (Reflects 95th percentile w/o CHF ):
  18-<44 yr: 36-178 pg/mL 44-<54 yr: 36-192 pg/mL 54-<64 yr: 36-226 pg/mL 64-<74 yr: 36-353 pg/mL >74 yr: 36-624 pg/mL
Time Frame: Baseline and weeks 4 (+/- 3 days), 12 (+/- 3 days), and 24 (+/- 7 days)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
Number analyzed (Participants) | 10 | 6
pg/ml
  Baseline | 1070 (1310) | 666 (283)
  Week 4 | 1160 (1300) | 900 (402)
  Week 12 | 1310 (1270) | 633 (714)
  Week 24 | 846 (506) | 367 (366)
Statistical Analysis 1: Comparison: Experimental Treatment Oral Hymecromone (H01) vs Placebo; There is no significant difference in the mean secondary endpoint (NT-proBNP) at 24 weeks between the treatment (H01) and placebo group; Test type: Superiority; p = 0.442, Mixed Models Analysis; Mean Difference (Final Values) = 231.47, 95% CI 2-sided [-377.26 to 840.20]

9. Other Pre Specified Outcome: Inflammatory Markers and PH-specific Biomarkers (ESR, HSCRP)
Description: Change in inflammatory markers and PH-specific biomarkers (ESR, HSCRP)
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Pro-inflammatory Cytokines
Description: Change in pro-inflammatory cytokines
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: Change in Forced Expiratory Volume in one second (FEV1)
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Forced Vital Capacity (FVC) From Pulmonary Function Test (PFT)
Description: Change in Forced Vital Capacity (FVC) from pulmonary function test (PFT)
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Total Lung Capacity (TLC) From Pulmonary Function Test (PFT)
Description: Change in Total Lung Capacity (TLC) from pulmonary function test (PFT)
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Lung Diffusion Capacity (DLCO) From Pulmonary Function Test (PFT)
Description: Change in Lung diffusion capacity (DLCO) from pulmonary function test (PFT)
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exhaled Breath Condensate (EBC) Hyaluronan Concentrations
Description: Change in exhaled breath condensate (EBC) hyaluronan concentrations
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Pharmacokinetics (H01 and Metabolite Serum Concentrations)
Description: Describe the pharmacokinetics (H01 and metabolite serum concentrations)
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: HA Fragment Size
Description: Describe HA fragment size
Time Frame: Baseline to end of treatment (Week 24)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Experimental Treatment Oral Hymecromone (H01) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/6
Other Adverse Events (participants affected / at risk) | 3/10 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Treatment Oral Hymecromone (H01) (N=10) | Placebo (N=6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Not Related
Thromboembolic event (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not Related
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not Related
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Treatment Oral Hymecromone (H01) (N=10) | Placebo (N=6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 — Not Related
Lung infection (Infections and infestations) | 2 | 0 — Not Related
Fatigue (General disorders) | 0 | 1 — Possibly Related
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Not Related
Creatinine increased (Investigations) | 0 | 1 — Not Related
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Possibly Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05128929/Prot_SAP_000.pdf